CLINICAL TRIAL: NCT02962544
Title: Comparison Between Femtosecond Assisted LASIK and Small Incision Lenticule Extraction (SMILE) for Correction of Myopia and Myopic Astigmatism
Brief Title: Comparison Between FS- LASIK and FS-SMILE for Correction of Myopia and Myopic Astigmatism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Adel Mohamed El-mayah, Assistant lecturer, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151
Record Dates: First submitted 2016-10-24; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Myopia
Keywords: Femtosecond; Small incision lenticule extraction; Lenticule extraction; LASIK; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visumax device for FS-SMILE group (Active Comparator): (FS-SMILE )femtosecond small incision lenticule extraction procedure using Visumax laser device as a surgical intervention for correction of myopia and myopic astigmatism will be done for 30 eyes of patients with myopia or myopic astigmatism.
  Interventions: Procedure: FS-SMILE; Device: Visumax device
- FS 200 device for FS-LASIK group (Active Comparator): (FS-LASIK)femtosecond assisted LASIK procedure using Fs200 laser device as a surgical intervention for correction of myopia and myopic astigmatism will be done for 30 eyes of patients with myopia or myopic astigmatism.
  Interventions: Procedure: FS- LASIK; Device: FS 200 device

INTERVENTIONS:
Procedure: FS-SMILE — The procedure will be performed using an established technique. the patient's eye will be centered and docked with the curved interface cone before application of suction fixation.The laser will be activated for photo-dissection in the following sequence: first the posterior surface of the refractive lenticule then the lenticule border then The anterior surface of the refractive lenticule which extended beyond the posterior lenticule diameter by 0.5 mm to form the anterior flap and is followed by a rim cut. After the suction is released, a Siebel spatula is inserted under the cap near the hinge before the cap is separated. The edge of the refractive lenticule is separated from the stromal bed with a sinsky hook and the posterior border of the lenticule gently separated with the Siebel spatula. The lenticule is then grasped with forceps through the small incision.
  Arms: Visumax device for FS-SMILE group
Procedure: FS- LASIK — LASIK procedure Each LASIK procedure will be performed using a standard, established technique. Under topical anesthesia and standard draping, a lid speculum is used to retract the eyelids. A superiorly hinged 100 μm thick flap will be created using the WaveLight FS200 (Alcon Laboratories, Inc.) With inverted side cut (115 ̊) .Excimer laser ablation is then performed using WaveLight EX500 excimer laser (Alcon Laboratories, Inc.).After ablation, the flap will be carefully repositioned, and postoperative medications are commenced.
  Arms: FS 200 device for FS-LASIK group
Device: Visumax device
  Arms: Visumax device for FS-SMILE group
Device: FS 200 device
  Arms: FS 200 device for FS-LASIK group

SUMMARY:
Aim of the work is to compare the results of femtosecond assisted LASIK and small incision lenticule extraction (SMILE) as regards safety, efficacy and predictability. As a secondary outcomes , the investigators will compare the results of both techniques on corneal biomechanics, dry eye measures, corneal asphericity and higher order aberration.

DETAILED DESCRIPTION:
Rationale and Background

LASIK (laser in situ keratomileusis) is a surgical procedure designed to correct refractive errors. LASIK involves creating a corneal flap using a microkeratome followed by reshaping the cornea using an excimer laser to remove tissue from the underlying stromal bed and then replacing the corneal flap.

LASIK evolved from a variety of techniques in refractive surgery. Keratomileusis, with both freeze and non-freeze techniques was used in the USA in the 1970s.This procedure was followed by automated lamellar keratoplasty (ALK), in which a microkeratome was used to create either a free cap or a hinged corneal flap. Tissue from the corneal bed was removed to alter the refractive error and the flap was replaced. Keratomileusis and ALK were relatively imprecise mechanical techniques. After the ophthalmic excimer laser has been developed, it has been used to reshape the cornea in a technique called photorefractive keratectomy (PRK). LASIK combines the technique of creating a hinged corneal flap from ALK with excimer laser ablation from PRK. Potential advantages of LASIK over PRK include earlier postoperative stabilization and faster improvement of visual acuity, less postoperative patient discomfort, shorter duration of postoperative medication use and an easier enhancement procedure.

However LASIK -like any other surgical procedures- is not without complications. Complications of LASIK include dry eye, glare and night vision complaints and the most serious flap complications which include button hole, free cap, incomplete flap, infection and inflammation.

Femtosecond lasers have been widely used in LASIK to fashion a corneal flap instead of mechanical microkeratome, which is followed by corneal ablation using excimer laser. The advantages of femotosecond or 'bladeless' LASIK over microkeratome LASIK flaps are more precise flap thickness, reduced postoperative dry eye symptoms, reduced flap dislocation and reduced incidence of buttonholes or free caps.

Recently, refractive lenticule extraction (ReLEx) has been introduced as a single laser refractive procedure (all-in-one femtosecond LASIK) without the use of an excimer laser. Small incision lenticule extraction (SMILE) is a variation of ReLEx which requires no retractable flap so reducing the incidence of flap complications, dry eye, reducing the surgical time and patient discomfort through operating on only one device in addition to decreasing the risk of ectasia.

Patients and methods Type of study Our study is a prospective, non-randomized, comparative clinical study applied on patients with myopia or myopic astigmatism.

Treatment group The study will include 60 eyes of patients with myopia or myopic astigmatism presenting for refractive correction. Femtosecond assisted LASIK group will include 30 eyes and SMILE group will include 30 eyes.

Pre-operative examination

All patients will undergo complete ophthalmological examination before surgery, including:

* Uncorrected and best corrected visual acuity assessement using snellen visual acuity chart.
* Manifest refraction.
* Slit lamp examination.
* IOP measurement.
* Dilated fundus examination
* Assessment for dry eye using Schirmer test and tear break up time test (TBUT).
* Corneal topographic analysis using combined Schimpflug and placido disc imaging principles using CSO topography system (CSO, Firenze, Italy).
* Wavefront analysis.
* Corneal biomechanical parameters using Ocular Response Analyzer (ORA; Reichert Inc, Depew, NY).

Surgical procedure LASIK procedure Each LASIK procedure will be performed using a standard, established technique. Under topical anesthesia and standard draping, a lid speculum is used to retract the eyelids. A superiorly hinged 100 μm thick flap will be created using the WaveLight FS200 (Alcon Laboratories, Inc.) With inverted side cut (115 ̊) .Excimer laser ablation is then performed using WaveLight EX500 excimer laser (Alcon Laboratories, Inc.).After ablation, the flap will be carefully repositioned, and postoperative medications are commenced.

SMILE procedure Each SMILE procedure will be performed using an established, described technique. After application of topical anesthesia, standard sterile draping, and insertion of the speculum, the patient's eye will be centered and docked with the curved interface cone before application of suction fixation.

The laser will be activated for photo-dissection in the following sequence: first the posterior surface of the refractive lenticule (spiral in), then the lenticule border is created. The anterior surface of the refractive lenticule (spiral out) is then formed which extended beyond the posterior lenticule diameter by 0.5 mm to form the anterior flap and is followed by a rim cut.

After the suction is released, a Siebel spatula (Rhein Medical, Heidelberg, Germany) is inserted under the cap near the hinge before the cap is separated. The edge of the refractive lenticule is separated from the stromal bed with a sinsky hook and the posterior border of the lenticule gently separated with the Siebel spatula. The lenticule is then grasped with non-toothed serrated forceps through the small incision.

Postoperative management

Postoperative treatment:

* Topical tobramycin and dexamethasone eye drops (Tobradex; Alcon Laboratories, Inc., Fort Worth, TX) was used postoperatively every 6 hours for 1 week and stopped.
* Topical lubricants was also prescribed to be applied every 6 hours for 1 month (refresh liquigel, Allergan Laboratories, Inc.).

Postoperative assessment:

• Postoperative visits were scheduled for the first postoperative day, 1 month and 3 months after surgery. On the first postoperative day, UCVA measurement and slit-lamp examination (flap position and corneal integrity) will be performed. Three months after surgery, the same clinical examinations as preoperatively was performed.

Statistical analysis Data will be presented in terms of parametric and non-parametric data. Parametric data will be analyzed with paired student t test. Non-parametric data will be analyzed with Wilcoxon test. Statistical significance will be considered at 95% confidence interval. All tests will be two tailed and considered significant at p < 0.05 and highly significant at p < 0.01.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18 years or older.
2. Best corrected visual acuity of 6/6.
3. Manifest refraction spherical equivalent (MRSE) not more than 9diopters (D).
4. Refractive cylinder not more than 3 diopters (D).
5. No topographic evidence of forme frust keratoconus (FFKC).
6. No progressive change of sphere or cylinder more than 0.5 diopter per year.

Exclusion Criteria:

1. Previous history of ocular trauma or ocular surgery.
2. Concomitant active or previous ocular disease such as uveitis and glaucoma.
3. Systemic diseases affecting wound healing such as diabetes mellitus, collagen vascular diseases
4. Dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
refractive predictability(manifest refraction spherical equivalent using autorefractometer) | change from baseline at 3 months postoperative.
  • Refractive predictability, which is defined as the proportion number of eyes achieving a postoperative spherical equivalent (SE) within ±0.50 D of the intended target.
efficacy(Unaided distance visual acuity using snellen chart) | change from baseline at 3 months postoperative.
  Efficacy: defined as the proportion number of eyes achieving an unaided visual acuity (UDVA) of 20/20 or better postoperatively (efficacy= postoperative UCVA/preoperative BCVA %).
safety( Corrected distance visual acuity using snellen chart) | change from baseline at 3 months postoperative.
  Safety: defined as the proportion number of eyes that lost or gained one or more lines of postoperative best corrected visual acuity (BCVA) relative to the preoperative BCVA (Safety= Postoperative BCVA/preoperative BCVA %)

SECONDARY OUTCOMES:
corneal hysteresis | change from baseline at 3 months postoperative.
  corneal hysteresis will be measured by ORA device and the investigators will compare between the preoperative and postoperative results in both groups.
schirmer test | change from baseline at 3 months postoperative.
  schirmer test and tear breack up time test will be tested pre and postoperatively and the investigators will compare between the preoperative and postoperative results in both groups.
corneal higher order aberrations.( total RMS) | change from baseline at 3 months postoperative.
  corneal higher order aberrations( total RMS) will be measured and comparison between the preoperative and postoperative value will be conducted.
corneal resistance factor | change from baseline at 3 months postoperative.
  corneal resistance factor will be measured by ORA device and the investigators will compare between the preoperative and postoperative results in both groups.
tear break up time test. | change from baseline at 3 months postoperative.
  tear breack up time test will be tested pre and postoperatively and the investigators will compare between the preoperative and postoperative results in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen N Salem, MD, Study Director — Kasr alainy school of medicine; mohamed H hosny, MD, Study Director — Kasr alainy school of medicine; MOHAMED ANIS, MD, Study Director — Kasr alainy school of medicine
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No